CLINICAL TRIAL: NCT01063712
Title: Safety and Effectiveness of the Device "Nit-Occlud® PDA-R" for Percutaneous Closure of Patent Arterial Duct Between 2 and 8 mm in Patients Treated Interventionally in Specialized Centers
Brief Title: Safety and Effectiveness of the Device "Nit-Occlud® PDA-R"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pfm S.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFM-P034; Bioethics Committee (Registry Identifier: 08-06-2009)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Congenital Heart Disease
Keywords: Ductus; Patent ductus Arterious; "Nit-Occlud® PDA-R"; Interventional closure of PDA; Percutaneous closure
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nit-Occlud PDA-R (Other): Interventional, prospective clinical study, non randomized.
  Interventions: Device: Nit-Occlud® PDA-R

INTERVENTIONS:
Device: Nit-Occlud® PDA-R — Transcatheter implantation of a PDA Device (Nitinol) The catheterism was done under sedation, using a protocol established by inserting a catheter through a femoral artery and/or vein directed to the heart and great vessels. Invasive measurements are obtained in the descending aorta and pulmonary artery. Once in ductal position, we inject iodinated contrast medium that allows us to observe via X-ray the ductal morphology; obtaining accurate measurements to choose the appropriate device. The device is then inserted via the catheter, closing the ductus.
  The catheterism provides measures of aortic and pulmonary pressure, before, during and after the closure.
  Other Names: Device - Med - Nit Occlud PDA

SUMMARY:
The purpose of this study is to evaluate the safety and the effectiveness of the device "Nit-Occlud® PDA-R" in the percutaneous closure of patent ductus.

DETAILED DESCRIPTION:
During the years 2003 to 2008, the Cardiological Medical Center "Kardiozentrum" evaluated 1136 patients with echocardiographic studies, 14.7% of the patients were diagnosed with patent arterial duct. The PDA is an abnormal communication between the aorta and pulmonary artery. Untreated it can rise the intrapulmonary pressure and lead to serious complications like cardiac insufficiency.

The incidence of ducts as an isolated heart disease is between 3.6 and 7% of all congenital heart diseases at sea level, and 10 - 14% at high altitude; rising up to 20% in cities at more than 2.500 m about sea level. The ducts at high altitude are generally wider and larger than at sea level.

One treatment alternative is a percutaneous transluminal implantation of a permanent implant which closes the defect. The device under investigation "Nit-Occlud® PDA-R" is developed for closure of the PDA with a minimal diameter of 2-8 mm.

The device performs the function of generating the defect occlusion by the body itself. The implant stimulates the body to generate an epithelium over the implant so that the PDA closes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and echocardiographic compatibility with PDA without associated heart disease requiring surgical solution
* Minimum diameter of the PDA 2 to 8 mm
* Systolic pulmonary pressure measured during cardiac catheterization, not on pass 2/3 of the values of the systolic systemic pressure
* Weight higher than 10 kg, regardless of age
* Patients who were diagnosed and recruited during the period 2009 - 2010
* Patients with trisomy 21 also fulfill the previous criteria, the number of patients with T21 will not exceed 10% of the entire group of patients.
* letter of consent signed by parents or legal guardian

Relative Exclusion Criteria:

* Infections that occur during acute bacteremia, viremia, which can be treated
* Febrile syndrome
* Tooth decay
* Once the acute solved considering the patient's inclusion into the study

Exclusion Criteria:

* Pregnant women
* Pulmonary hypertension, increased to 2 / 3 of systemic pressure
* Eisenmenger syndrome
* Other associated heart disease, requiring surgical solution
* Immuno-compromised patients
* Pathology oncology
* Hematologic or coagulation disorders
* Allergy to contrast medium
* Atypical or calcified Ductus
* Parents or legal guardians who do not accept the risks of catheterization
* Parents or legal guardians and patients who do not accept to sign the letter of consent or who revoke the consent.
* Patients who participated in another clinical investigation during the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Heath, MD, Ph.D, Principal Investigator — Kardiozentrum
Locations (1):
- Kardiozentrum and Surgical Medical Center Boliviano Belga, La Paz, Murillo, Bolivia

REFERENCES:
- [Background] Lang N, Schmitz C, Lehner A, Fuchs F, Heath A, Freudenthal F, Wintersperger BJ, Huber AM, Thein E, Netz H, Kozlik-Feldmann R. Preclinical evaluation of a new self-expanding device for closure of muscular ventricular septal defects in a pig model. Catheter Cardiovasc Interv. 2010 Feb 15;75(3):408-15. doi: 10.1002/ccd.22285. PMID 19882712
- [Background] Heath A, Lang N, Levi DS, Granja M, Villanueva J, Navarro J, Echazu G, Kozlik-Feldmann R, del Nido P, Freudenthal F. Transcatheter closure of large patent ductus arteriosus at high altitude with a novel nitinol device. Catheter Cardiovasc Interv. 2012 Feb 15;79(3):399-407. doi: 10.1002/ccd.23302. Epub 2011 Dec 12. PMID 21805617
- [Result] Freudenthal FP, Heath A, Villanueva J, Mendes J, Vicente X, von Alvensleben I, Echazu G, Navarro J, Lang N, Kozlik-Feldmann R. Chronic hypobaric hypoxia, patent arterial duct and a new interventional technique to close it. Cardiol Young. 2012 Apr;22(2):128-35. doi: 10.1017/S1047951111000990. Epub 2011 Jul 21. PMID 21774843
- See also: CSI Frankfurt 08´ - Closure of Very Large PDAs with New Device — http://www.csi-congress.org/index.php?=812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective clinical study between June 2009 and December 2010 in La Paz, Bolivia. 29 out of 59 patients selected with inclusion and exclusion criteria(≥ 10 Kg, Patient Arterial Duct of 2 - 8 mm minimal diameter, "Nit-Occlud® PDA-R" used, systolic pulmonary pressure ≤ 67% of systolic aortic pressure and absence of any other chronic disease).
Pre-assignment Details: 30 patients were excluded. Four and eight patients with Patent Arterial Duct bigger than 8 mm or smaller than 2 mm, eleven patients with pulmonary pressure elevated more than 67% of systolic pressure, nine patients lighter than 10 Kg and three patients with atypical ducts. Some were excluded for more than one reason.
Groups:
- "Nit-Occlud® PDA-R" Implantations Group: Children born with patent arterial duct develop cardiac insufficiency early in life, show failure to thrive and frequent respiratory infections. Pulmonary hyperflow through the duct can lead to changes in the pulmonary vasculature and irreversible pulmonary hypertension. This can be prevented if we close the ducts on time. The classical method is open thorax surgery, which involves deep anaesthesia, a scar, possible complications (thorax deformities and instability) and a long stay in hospital. With the Interventional Closure of Patent Arterial Duct technique the patients stay only one day in hospital, the thorax is not open, and only slight sedation is needed. The device closure and the surgery have similar closure rates, but there are fewer complications using the intervention method, and it is also less expensive.
  This group of patients were chosen because they have ducts in mean sizes (2-8 mm), haven´t developed pulmonary hypertension and have enough weight to be treated.
Period: Overall Study
Arm/Group | "Nit-Occlud® PDA-R" Implantations Group
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Effectiveness of the Device: "Nit-Occlud® PDA-R": Children born with patent arterial duct develop cardiac insufficiency early in life, show failure to thrive and frequent respiratory infections. Pulmonary hyperflow through the duct can lead to changes in the pulmonary vasculature and irreversible pulmonary hypertension. This can be prevented if we close the ducts on time. The classical method is open thorax surgery, which involves deep anaesthesia, a scar, possible complications (thorax deformities and instability) and a long stay in hospital. With the Interventional Closure of Patent Arterial Duct technique the patients stay only one day in hospital, the thorax is not open, and only slight sedation is needed. The device closure and the surgery have similar closure rates, but there are fewer complications using the intervention method, and it is also less expensive.
  This group of patients were chosen because they have duct in mean sizes (2-8 mm), haven´t developed pulmonary hypertension and have enough weight to be treated.
Arm/Group | Effectiveness of the Device: "Nit-Occlud® PDA-R"
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 7
Region of Enrollment [Number; unit: units=participants]
  Bolivia | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Closed Patent Ductus Arteriosus (Defect) Determinated by Echocardiography ( Time Frame: One Year After Treatment)
Description: The closure rate is an effectiveness outcome. Complete closure without a residual shunt is defined as absence of color flow (an echocardiographic technique used to observe the flow of blood in the heart) between the aorta and the pulmonary artery through the duct. Additionally, the position of the device, regression of the dilation of the left ventricle and left atrium and assessing of unrestricted doppler flow in the descending aorta and left pulmonary artery were documented. Clinical status was also assessed.
Time Frame: up to one year after percutaneous closure
Population: 29 patients were controled in a period of one year and were examinated by echocardiography.The number of patients who showed no more duct bloodflow (seen with color doppler echocardiography or "color flow") in the control period is given as number and as percentage of the complete group.
Measure: Number; unit: Participants
Groups:
- Closure in the Control Period: The number of patients who showed no more duct bloodflow (seen with color doppler echocardiography or "color flow") in the control period is given as number and as percentage of the complete group.
Arm/Group | Closure in the Control Period
Number analyzed (Participants) | 29
Participants
  Complete closure at time 1 (immediate) | 19
  Complete closure at time 2 (24 hours) | 23
  Complete closure at time 3 (1 month) | 28
  Complete closure at time 4 (3 months) | 29
  Complete closure at time 5 (6 months) | 29
  complete closure at time 6 (12 months) | 29
  partially open at time 1 (immediate) | 10
  partially open at time 2 (24 hours) | 6
  partially open at time 3 (1 month) | 1
  partially open at time 4 (3 months) | 0
  partially open at time 5 (6 months) | 0
  partially open at time 6 (12 months) | 0
Statistical Analysis 1: Comparison: Closure in the Control Period; It is not a analysis of two groups. Only one group of patients was analyzed; Test type: Superiority or Other; p < 0.01, percentage

2. Secondary Outcome: Number of Patients With a Decreased Dilation of the Left Heart Chamber (Time Frame: One Year After Treatment). Dilation of the Left Ventricle and Left Atrium Was Measured Before and One Year After Implantation by Echocardiography.
Description: The patients were examined clinically and echocardiographically after 24 hours, one month, three months and six months after the percutaneous closure. Dilation of the left ventricle and left atrium are consequences of the hyperflow through the ducts. Regression of both ventricle and atrium are expected after closure of the ducts and can be documented by echocardiography. Additionally, the position of the device and the doppler flow in the descending aorta and left pulmonary artery were documented.
Time Frame: one year after percutaneous closure
Population: The patient selection was based in the "consecutive case" and "intention to treat" method. All patients recruited in the determinated time frame (June 2009 to May 2010) who met the initial inclusion criteria were treated in the catheterisation laboratory. There the definite inclusion criteria were applied.
Measure: Number; unit: participants
Groups:
- Number of Patients With Complete Regression of Dilation: Children born with patent arterial duct develop cardiac insufficiency early in life. Pulmonary hyperflow through the duct can lead to changes in the pulmonary vasculature and irreversible pulmonary hypertension. This can be prevented if we close the duct on time. The device closure and the surgery have similar closure rates, but there are fewer complications using the intervention method.
  This group of patients had 2-8 mm ductus, haven´t developed pulmonary hypertension and have enough weight to be treated.
  Patients with left to right shunt show a dilation of left ventricle and left atrium. The quotient Left atrium/aortic ring is a well known method to estimate the grade of the dilation of the left atrium. The M-Mode method, is useful to assessed the regression of the ventricle after the ducts is closed. These observations were made at the beginning of the study and after six months.
Arm/Group | Number of Patients With Complete Regression of Dilation
Number analyzed (Participants) | 29
participants
  Regression at time 1 (immediate) | 29
  Regression at time 5 (6 months) | 29
Statistical Analysis 1: Comparison: Number of Patients With Complete Regression of Dilation; It is a one arm clinical study. No comparison between groups was made; Test type: Superiority or Other; p < 0.01, percentage; The analysis was made on the basis of the percentage of patients with completely regressed dilation

ADVERSE EVENTS:
Time Frame: Data on adverse effects was collected over 18 months. Clinical, laboratory and echocardiographic findings were documented in a established protocol.
Description: Controls were made at 24 hours, one week, 1 month, 3 months, six months and 1 year.
Arm/Group | Effectiveness of the Device: "Nit-Occlud® PDA-R"
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
The number of participants is small, because the participants were recruited in high altitude cities over 2700m above the sea level. At this altitude bigger defects are more frequent to find than little ones, so is pulmonary hypertension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No